CLINICAL TRIAL: NCT03955601
Title: A Novel TBI Free Conditioning Protocol for Haploidentical Hematopoeitic Stem Cell Transplant in Acquired Aplastic Anemia
Brief Title: A Novel TBI Free Conditioning Protocol for Haploidentical Transplant in Acquired Aplastic Anemia:
Acronym: FluCAB-Prime
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFBMTC-HAPLO-AA
Record Dates: First submitted 2019-04-22; First posted 2019-05-20 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Aplastic Anemia Idiopathic
Keywords: haploidentical; Aplastic anemia; TBI
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TBI free Haploidentical HSCT (Experimental): Recipients will receive a reduced intensity conditioning regimen of ''Fludarabine'' 30 mg/m2 IV daily from day -7 to -3, ''Cyclophosphamide'' 14.5-30 mg/kg IV daily on day -6 and -5 , ''rabbit Antithymocyte globulin'' 5 mg /kg/day from day -6 to day-3; ''Busulphan'' IV 3.2 mg per kg/day in 02 divided doses on day -3 and day-2, ''Granulocyte Colony Stimulating factor primed Bone marrow harvest'' and/OR ''PBSC'' graft on day 0 and day +1 respectively and Graft versus host disease prophylaxis with ''post-transplant cyclophosphamide'' administered at a dose of 50mg/kg/day given daily on days +3 and +5 post-transplant and ''cyclosporine'' from day +5, ''mycophenolate mofetil'' from day+5 to day+35.
  Interventions: Drug: Haploidentical HSCT using TBI free regimen, ''ATG'' with ''Post transplant cyclophosphamide''

INTERVENTIONS:
Drug: Haploidentical HSCT using TBI free regimen, ''ATG'' with ''Post transplant cyclophosphamide'' — ''Busulphan'' will be used in place of ''TBI'' in equivalent myelotoxic dose to facilitate engraftment , ''ATG'' will be used to reduce GVHD and facilitate engraftment while ''combine PBSC'' and/OR ''Bone marrow harvest'' will be used
  Other Names: ''Combined BMH'' and ''PBSC harvest''

SUMMARY:
Severe and very severe aplastic anemia are life threatening disorders for which allogeneic stem cell transplant is only curative treatment. However, matched sibling donor (MSD) is available in only 25-35% cases. Pakistan has a population of around 203 million but there is no donor registry available so there is no option available for matched unrelated donor (MUD) transplants . Haploidentical transplant represents only curative option for patients lacking MSD. Protocols involving post transplant cyclophosphamide require Total body irradiation (TBI) and utilize peripheral blood stem cell(PBSC) as graft source. TBI is not available in most of transplant centres across Pakistan due to lack of availability , cost and lack of expertise. The investigators have conceived a novel TBI free conditioning regimen to be used for haplo-identical Hemtopoeitic stem cell transplant in acquired aplastic anemia patients

DETAILED DESCRIPTION:
Aplastic anemia is considered to be a rare and heterogenous disease with incidence of 1-2 per million in western countries. Data from Asian studies show a 3-4 fold higher incidence.Majority of newly diagnosed aplastic anemia patients are younger and in Armed forces bone marrow transplant cohort of 1324 patients 64 % patient are younger than 24 years of age and 87% patients younger than 40 years (unpublished data).There is no donor registry in Pakistan and patients lacking sibling match donor cannot proceed to stem cell transplant due lack of matched unrelated donors. Horse antithymocyte globulin is not available currently in Pakistan and response to Rabbit antithymocyte globulin is dismal as shown in number of international studies. So haploidentical stem cell transplant remains only curative option for patients lacking Matched sibling donor. Currently there are 2 major platforms used for haplo-identical stem cell transplant. Post transplant cyclophosphamide based using TBI and haplo regimen of Peking university. TBI is not available for most of our patients in Pakistan due to cost,non-availability and lack of expertise. The investigators have formulated a novel TBI free regimen incorporating Busulphan, antithymocyte globulin and using co-primed bone marrow and peripheral blood harvest to minimize graft-versus-host disease and facilitate engraftment. Post transplant cyclophosphamide, Cyclosporine and mycophenolate mofetil will be used for graft-versus-host disease prophylaxis

ELIGIBILITY:
Inclusion Criteria:

* Age >2 years and < 60 years
* Karnofsky performance status >= 70%
* Aplastic Anemia that meets the following criteria:

  i. Peripheral Blood (must fulfill 2 of 3): ii. <500 neutrophils iii. <20,000 platelets iv. absolute reticulocyte count <40,000/microL
* Bone Marrow (must be ): markedly hypocellular (<25% of normal cellularity) with absence of reticulin and abnormal infiltrate

Exclusion Criteria:

* Presence of donor specific antibodies
* Fanconi anemia
* Cytogenetic abnormalities suggestive of myelodysplastic syndrome
* Prior HSCT
* Human immunodeficiency virus infection
* Active Hepatitis B virus infection
* Active /uncontrolled bacterial, viral , fungal infection or Tuberculosis
* Psychiatric illness
* Poor cardiac function (ejection fraction <40%)
* Poor pulmonary function (Forced vital capacity <50% predicted)
* Poor liver function (bilirubin >= 2mg/dL)
* Poor renal function (creatinine >= 2.0mg/dL or creatinine clearance <40)

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with overall survival | from the date of transplant to 1 year post transplant
  overall survival is defined as the time interval from date of transplant to death or to last follow-up, whichever occurs first.

SECONDARY OUTCOMES:
Number of Participants with Disease free survival | from the date of transplant to 1 year post transplant
  from time of transplant to death or last follow up
Time of Neutrophil engraftment | from the date of transplant to 10 to day 28 post transplant
  first of 3 consecutive days with Absolute neutrophil count> 0.5
Frequency of Graft versus host disease | from the date of transplant to acute upto 100 day post transplant, chronic >100 days post transplant
  as per clinical and histopathological diagnosis
Rate of Complications | from the date of transplant to 1 year from day of transplantation
  both infectious and non infectious

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Mehmood Satti, FCPS, Study Chair — NIBMT
Locations (1):
- NIBMT, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No